CLINICAL TRIAL: NCT00935649
Title: Multi-Center Trial: Evaluation of PinPointe FootLaser Treatment for Infected Toenails (Onychomycosis)
Brief Title: PinPointe FootLaser for the Treatment of Onychomycosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PathoLase, Inc. (Industry)
Responsible Party: David M Harris, PhD, PathoLase, Inc
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CLN0001.p.A
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2010-11

CONDITIONS: Infected Toenails; Onychomycosis
Keywords: Toenail Fungus; PinPointe; FootLaser; Onychomycosis; Fungal nails
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Randomized great toe (Experimental): Subjects with both great toes infected. Right/left randomized to treatment / no treatment
  Interventions: Device: PinPointe FootLaser
- Untreated Toe (No Intervention)

INTERVENTIONS:
Device: PinPointe FootLaser — Medical laser
  Arms: Randomized great toe

SUMMARY:
To evaluate the safety and efficacy of the PathoLase FootLaser treatment of infected toenails.

DETAILED DESCRIPTION:
The study is a multi-center controlled study evaluating laser treatments of infected great toes in a randomized blinded study of approximately 125 subjects. Right and left great toes are randomized to treatment or no treatment. Samples from infected areas are sampled and evaluated for presence of fungus with KOH, PCR and culture tests. Nail bed clearing and nail plate growth are measured from high resolution photographs by a blinded evaluator. Subjects will be evaluated at baseline and at 8, 16, 24 and 48 weeks for safety and effectiveness of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of either sex,
* 18-80 years of age,
* Both great toes with clinical signs of infection.
* Positive KOH or culture test

Exclusion Criteria:

* Existing or history of cancer/skin malignancy,
* Use of oral antifungal agents in past 6 months,
* Use of topical antifungal agents in past 1 month,
* Loss of protective sensation in either foot,
* Infection involving lunula of either great toe,
* Longitudinal streaks/spikes of either great toenail,
* Distal nail thickness > 2 mm of either great toe,
* Prior surgical treatment of either great toe in past 12 months,
* Participation in another medical device/pharmaceutical study,
* Condition that investigator determines makes it unsafe for subject to participate,
* Pregnancy, breastfeeding or plans to become pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Harris, PhD, Study Director — PathoLase, Inc.; Bernard Goffe, MD, Principal Investigator — Dermatology Associates
Locations (4):
- United States (3):
  - Rochester Laser Center, Rochester, New York
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Dermatology Associates, Seattle, Washington
- Mediprobe Research Inc, London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Randomized Great Toe
Started | 139
Completed | 134
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Randomized Great Toe
Number analyzed (Participants) | 139
Age Continuous [Mean (Standard Deviation); unit: years] | 52.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 101

OUTCOME MEASURES:

1. Primary Outcome: Nail Bed Clearing
Description: Change in amount of clear nail over time.
Time Frame: 48 weeks
Population: There was a fatal design flaw to the trial. We were advised to collect nail samples for mycologic analysis at every visit. As a result investigators were removing our primary outcome variable, increase in clear nail, at each visit. Consequently our estimates of nail growth following treatment are inaccurate and invalid.
Groups:
- Treated Great Toe: Laser treatment of great toe
- Untreated Great Toe: untreated control great toe
Arm/Group | Treated Great Toe | Untreated Great Toe
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mycology
Description: KOH, PCR and cultures of patients who were bilaterally positive or negative for each test.
Time Frame: 48 weeks
Population: as for outcome 1
Arm/Group | Treated Great Toe | Untreated Great Toe
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: Adverse events not assessed for untreated toe. Adverse events are per toe not per patient.
Arm/Group | Treated Great Toe | Untreated Great Toe
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/0
Other Adverse Events (participants affected / at risk) | 15/139 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treated Great Toe (N=139) | Untreated Great Toe (N=0)
intraoperative foot pain (Surgical and medical procedures) | 15 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes